CLINICAL TRIAL: NCT03242291
Title: Evaluation of Marginal Integrity of Hydroxyapatite Nano-Fiber Reinforced Flowable Composite Versus Conventional Resin-Based Flowable Composite in Initially Demineralized Pits and Fissure: A One Year, Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, donia elshafey, internal resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEBC-CU-2017-7-29
Record Dates: First submitted 2017-07-31; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Marginal Integrity of Hydroxyapatite Nanofiber Reinforced Flowable Composite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional resin-based flowable composite (Active Comparator)
  Interventions: Other: Conventional resin-based flowable composite; Other: Hydroxyapatite Nanofiber reinforced flowable composite
- Hydroxyapatite Nanofiber reinforced flowable composite (Other)
  Interventions: Other: Conventional resin-based flowable composite; Other: Hydroxyapatite Nanofiber reinforced flowable composite

INTERVENTIONS:
Other: Conventional resin-based flowable composite — assessment of marginal integrity of Conventional resin-based flowable composite
Other: Hydroxyapatite Nanofiber reinforced flowable composite — assessment of marginal integrity of Hydroxyapatite Nanofiber reinforced flowable composite

SUMMARY:
This study will be conducted to evaluate the Marginal integrity of Hydroxyapatite Nanofiber reinforced flowable composite compared to a conventional resin-based flowable composite during management of initial carious lesion in adult population over a one year period.

DETAILED DESCRIPTION:
A total of 26 volunteer patients with at least 2 non-cavitated molar teeth will be assigned in this study. Patients will be divided into two groups according to type of flowable composite (R) where groups R1 the pits and fissure will be sealed with Hydroxyapatite Nanofiber reinforced flowable composite while groups R2 the pits and fissure will be sealed with conventional resin-based flowable composite. Each restoration will be assessed after one week, six and twelve months Both materials will be applied according to manufacturer's instructions where teeth should be cleaned to remove surface stains, then select appropriate shade of the flowable composite, A rubber dam is the preferred method of isolation, etch and rinse adhesive system is applied, where acid etching will be applied for 15 seconds then rinse and dry followed by application of adhesive then light cure 10 seconds, then place and cure in 2 mm increments of the flowable composite for 20 s., gently remove oxygen inhibition layer after light cure with slurry of pumice or polishing paste All restorations were reviewed after 1 week, 6, 12 months by two investigators who were blinded to the material used for the restorations. All restorations were be evaluated by calibrated examiners following the FDI criteria

ELIGIBILITY:
Inclusion Criteria:

* Patients should be over 18 Years old.
* Patient should have good oral hygiene and general health
* With at least 2 non-cavitated initial occlusal carious lesion first and/or Second molar teeth in each quadrant of maxilla or mandible

Exclusion Criteria:

* Known allergy to any of the resins used,
* Clinically detectable caries,
* Previously placed sealants or restorations,
* Bruxism or malocclusion

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
marginal integrity of both restorations | 12 months
  restorations will be reviewed after 12 months by two investigators who are blinded to the material used for the restorations. All restorations will be evaluated by calibrated examiners following the FDI criteria Data will be explored for normality using Kolmogrov-Smirnov test and Shapirowilk test. Comparisons between before and after treatment for normally distributed numeric variables will be done by Wilcoxon sign test. Comparisons between categorical variables will be performed using the chi square test Mcnemar test. A p-value less than or equal to 0.05 will be considered statistically significance. All tests will be two tailed.

IPD SHARING:
Plan to Share IPD: Undecided